CLINICAL TRIAL: NCT04749576
Title: Efficacy of Nutritional Saffron Supplement As An Anti Inflammatory Agent In Patients With Inflammatory Bowel Disease
Brief Title: Saffron as Anti Inflammatory Agent In Patients With Inflammatory Bowel Disease
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Howard University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HowardU
Record Dates: First submitted 2020-12-09; First posted 2021-02-11 (Actual); Last update posted 2021-02-11 (Actual); Status verified 2021-01

CONDITIONS: Ulcerative Colitis
MeSH Terms: conditions — Colitis, Ulcerative

STUDY DESIGN:
Intervention Model Description: randomize double placebo
Who Masked: Participant, Care Provider
Masking Description: Both patients and care provider does not know whether the participant receiving placebo or saffron
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Low dose saffron (Active Comparator): healthy, mild-moderate ulcerative colitis for low dose
  Interventions: Dietary Supplement: saffron supplement for IBD
- High dose Saffron (Active Comparator): healthy, mild-moderate ulcerative colitis for high dose
  Interventions: Dietary Supplement: saffron supplement for IBD
- Placebo (Placebo Comparator): healthy, mild-moderate ulcerative colitis for placebo
  Interventions: Dietary Supplement: saffron supplement for IBD

INTERVENTIONS:
Dietary Supplement: saffron supplement for IBD — anti inflammatory effect

SUMMARY:
Nutritional Saffron supplement has been widely used as food supplement and has known anti-depressant and anti-inflammatory activities. It is generally consumed as stigmas in drinks or dishes. The investigators use saffron extract in patients with colitis for 8 weeks.

DETAILED DESCRIPTION:
The patients invited to participate in a research study on Inflammatory Bowel Diseases (IBD) and saffron as a nutritional anti-inflammatory supplement.

Inflammatory Bowel Disease (IBD) is composed of Crohn's Disease (CD) and Ulcerative Colitis (UC). Continuous altered immune responses and inflammation associate with this disease. More than two-thirds of patients reported that IBD-associated symptoms negatively affected their quality of life and their performance at work.

* Patients with IBD are generally put on immunosuppressants (that block or slow participants' immune system to lower the level of inflammation). Long-term use of these immunosuppressants have some serious side effects.
* The goal of this protocol is to lower the need for these immunosuppressants by giving saffron as capsules in two different doses. The investigators will assess whether the addition of saffron will improve the overall patient's status and decrease the need for immunosuppressants. If participants have been prescribed immunosuppressants by the participant's doctor, saffron will be added to the participants' treatment.
* The investigators request that the subject answer as many questions as they can during this visit. If they are unable to complete the questionnaires during this visit, the investigators ask them to please return them within 7 days. If the investigators do not receive the questionnaires, the investigators will make one phone call to remind the subjects to send the questionnaires back.
* The subject medical record and colonoscopy report will be used to determine IBD or health status, the blood sample will be used to assess immune markers (inflammatory and antiinflammatory), stool sample will be used to assess some inflammation markers and saffron effect on the intestinal bacterial composition, a saliva sample will be used to assess whether saffron selectively affects the intestinal bacteria but not the saliva bacteria and the urine sample will be used to assess saffron release in body fluids.
* Participants are being asked to participate in this research project because participants are having a normal colonoscopy for screening, or IBD.
* If a biopsy is taken at colonoscopy. a pathologist will use a portion to make a diagnosis. The investigators are requesting permission to use a portion of the excess tissue that the pathologist does not need, for this research project.
* Samples will be collected at baseline (day 0) and 8 weeks later after saffron capsules utilization.
* This is a double-blind clinical trial, you will not know whether participants are given a placebo (capsule without saffron) or saffron dose 1 or 2. This is important for participants and for the study process, to avoid any psychological effect on the expected saffron effect.
* However, by the end of the 8 weeks and after collecting and analyzing the data from all participants, the investigators will inform the subject of what the subjects were given and potential next steps.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patients aged >18 years
2. Have UC diagnosed at least 3 months prior to screening? The diagnosis of UC must be confirmed by endoscopic and histologic evidence.
3. Men and women of childbearing potential must agree to use adequate birth control measures during the study.
4. Ability to provide written informed consent and to be compliant with the schedule of protocol assessments, treatment plan, laboratory tests, and other study procedures.
5. UC patients with mild, mod, severity as assess by the 4 scale assessment (Normal, mild, mod, severe).
6. Treatment naïve subjects diagnosed with ulcerative colitis (without previous exposure to treatment).

7. UC patients already on a treatment might be considered, with saffron as an add-on 8. UC patients who displayed no improvement with any available treatment might be considered for saffron as an alternative treatment in this option.

Exclusion Criteria:

1. Patients taking immunosuppressive medicine for a disease other than UC
2. Rheumatologic disease and other underlying diseases that can interfere with the study process.
3. Pregnancy
4. If the UC has been present for > 10 years, a colonoscopy with biopsy has to be performed to rule-out dysplasia.
5. A subject who had surgery as a treatment for ulcerative colitis or likely to require surgery during the study period.
6. Subjects with evidence of liver disease or abnormal liver enzymes and function tests (e.g. total bilirubin, aspartate aminotransferase (AST) or alanine aminotransferase (ALT) higher than the upper limit of normal) at the screening visit.
7. Subjects who have any condition possibly affecting oral nutritional supplement absorption.
8. Any other condition which in the opinion of the investigators would make the subject unsuitable for inclusion in the study.
9. Patients with known active or untreated GI infections including C. difficile, CMV, HSV, HIV

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2020-12-15 (Actual); Primary Completion 2021-12-10 (Estimated); Study Completion 2023-12-10 (Estimated)

PRIMARY OUTCOMES:
inflammatory markers assessment | 8 weeks
  Serum anti-inflammatory and pro-inflammatory markers measures in 8 weeks compared to baseline improving the blood immune marker in the normal range for contributing factors which consist of TNF-α (8.1 pg/mL).IL-1β (<5 pg/mL), IL-6(5-15 pg/ml)., and IL-10 (4.8-9.8 pg/ml), The units in the parenthesis are the normal range for each marker
stool frequency assessment | 8 week
  will be assessed by decreasing less than 2 per day
stool consistency assessment | 8 week
  Improvement to median score 4 to normal stool consistency. Bristol score: Improvement in stool consistency measures in 8 weeks in our study compared to baseline (Bristol score: The ideal stool is generally type 3 or 4, easy to pass without being too watery too solid. Type 1 or 2, it is sign of constipation. Types 5, 6, and 7 tend toward diarrhea)
fecal calprotectin assessment | 8 weeks
  Decrease in calprotectin levels. Fecal calprotectin normal range to be 10 to 60 μg/mg
C reactive protein assessment | 8 week
  change on C reactive protein level reading is less than 10 milligram per liter
erythrocyte sedimentation rate assessment | 8 weeks
  maintaining erythrocyte sedimentation rate with the normal range of 0 to 22 mm/hr for men and 0 to 29 mm/hr for women.
Serum Pro-inflammatory assessment | 8 weeks
  improving the blood immune marker in the normal range for contributing factors which consist of TNF-α (8.1 pg/mL).IL-1β (<5 pg/mL), IL-6(5-15 pg/ml)., IL-10 (4.8-9.8 pg/ml), and Th17 (221.6±90.2/µl). The units in the parenthesis are the normal range for each marker
Serum Anti-inflammatory assessment | 8 weeks
  improve the IL-10 level to at least reach the normal level of ranged from 4.8-9.8 pg/ml
The Ulcerative Colitis Colonoscopic Index of Severity scores | 8 weeks
  Decrease of 2 or more unit in the Ulcerative Colitis Colonoscopic Index of Severity score. The Ulcerative Colitis Colonoscopic Index of Severity scores for mild colitis is 3-5, and for moderate is 5-9

SECONDARY OUTCOMES:
endoscopy colitis assessment | 8-12 weeks
  Secondary endpoints will be endoscopy remission at week 8-12 according to gastroenterologist preference

CONTACTS AND LOCATIONS:
Overall Officials: Hassan Ashktorab, Study Chair — Howard Uinversity
Locations (1):
- Howard University Hospital, Washington D.C., District of Columbia, United States

IPD SHARING:
Plan to Share IPD: No
After completing the tials we will share the data

REFERENCES:
- [Result] 1 Ghosh S, Mitchell R. Impact of inflammatory bowel disease on quality of life: Results of the European Federation of Crohn's and Ulcerative Colitis Associations (EFCCA) patient survey J Crohns Colitis. 2007;1:10-20. 2 Jess T, Gamborg M, Munkholm P, Sorensen TI. Overall and cause-specific mortality in ulcerative colitis: meta-analysis of population-based inception cohort studies Am J Gastroenterol. 2007;102:609-617. 3 Tanaka T. Colorectal carcinogenesis: Review of human and experimental animal studies J Carcinog. 2009;8:5. 4 Torres J, Burisch J, Riddle M, Dubinsky M, Colombel JF. Preclinical disease and preventive strategies in IBD: perspectives, challenges and opportunities Gut. 2016;65:1061-1069. 5 Dahlhamer JM, Zammitti EP, Ward BW, Wheaton AG, Croft JB. Prevalence of Inflammatory Bowel Disease Among Adults Aged >/=18 Years - United States, 2015 MMWR Morb Mortal Wkly Rep. 2016;65:1166-1169. 6 Nguyen DL, Parekh N, Bechtold ML, Jamal MM. National Trends and In-Hospital Outcomes of Adult Patients With Inflammatory Bowel Disease Receiving Parenteral Nutrition Support JPEN J Parenter Enteral Nutr. 2016;40:412-416. 7 Kappelman MD, Rifas-Shiman SL, Porter CQet al. . Direct health care costs of Crohn's disease and ulcerative colitis in US children and adults Gastroenterology. 2008;135:1907-1913. 8 Blakeley-Ruiz JA, Erickson AR, Cantarel BLet al. . Metaproteomics reveals persistent and phylum-redundant metabolic functional stability in adult human gut microbiomes of Crohn's remission patients despite temporal variations in microbial taxa, genomes, and proteomes Microbiome. 2019;7:18. 9 Ashktorab H, Soleimani A, Singh Get al. . Saffron: The Golden Spice with Therapeutic Properties on Digestive Diseases Nutrients. 2019;11. 10 Mashmoul M, Azlan A, Khaza'ai H, Yusof BN, Noor SM. Saffron: A Natural Potent Antioxidant as a Promising Anti-Obesity Drug Antioxidants (Basel). 2013;2:293-308. 11 Hosseinzadeh H, Talebzadeh F. Anticonvulsant evaluation of safranal and crocin from Crocus sativus in mice Fitoterapia. 2005;76:722-724. 12 Hosseinzadeh H, Modaghegh MH, Saffari Z. Crocus sativus L. (Saffron) extract and its active constituents (crocin and safranal) on ischemia-reperfusion in rat skeletal muscle Evid Based Complement Alternat Med. 2009;6:343-350. 13 El-Maraghy SA, Rizk SM, Shahin NN. Gastroprotective effect of crocin in ethanol-induced gastric injury in rats Chem Biol Interact. 2015;229:26-35. 14 Hosseinzadeh H, Sadeghnia HR. Safranal, a constituent of Crocus sativus (saffron), attenuated cerebral ischemia induced oxidative damage in rat hippocampus J Pharm Pharm Sci. 2005;8:394-399. 15 Lee IA, Lee JH, Baek NI, Kim DH. Antihyperlipidemic effect of crocin isolated from the fructus of Gardenia jasminoides and its metabolite Crocetin Biol Pharm Bull. 2005;28:2106-2110. 16 Abdullaev FI, Espinosa-Aguirre JJ. Biomedical properties of saffron and its potential use in cancer therapy and chemoprevention trials Cancer Detect Prev. 2004;28:426-432. 17 Abdullaev FI. Cancer chemopreventive and tumoricidal properties of saffron (Crocus sativus L.) Exp Biol Med (Maywood). 2002;227:20-25. 18 Singh G, Brim H, Ashktorab H, Habtezion A. Protective effect of Saffron in mouse model colitis through immune modulation DDW Gasteroenrology, City;2020. 19 Yoshino F, Yoshida A, Umigai N, Kubo K, Lee MC. Crocetin reduces the oxidative stress induced reactive oxygen species in the stroke-prone spontaneously hypertensive rats (SHRSPs) brain J Clin Biochem Nutr. 2011;49:182-187. 20 Rahaiee S, Moini S, Hashemi M, Shojaosadati SA. Evaluation of antioxidant activities of bioactive compounds and various extracts obtained from saffron (Crocus sativus L.): a review J Food Sci Technol. 2015;52:1881-1888. 21 Hosseinzadeh H, Younesi HM. Antinociceptive and anti-inflammatory effects of Crocus sativus L. stigma and petal extracts in mice BMC Pharmacol. 2002;2:7. . 34 Maleki I, Taghvaei T, Barzin M, Amin K, Khalilian A. Validation of the Persian version of the inflammatory bowel disease questionnaire (IBDQ) in ulcerative colitis patients Caspian J Intern Med. 2015;6:20-24. 35 McGahuey CA, Gelenberg AJ, Laukes CAet al. . The Arizona Sexual Experience Scale (ASEX): reliability and validity J Sex Marital Ther. 2000;26:25-40. 36 Brim H, Yooseph S, Lee Eet al. . A Microbiomic Analysis in African Americans with Colonic Lesions Reveals Streptococcus sp.VT162 as a Marker of Neoplastic Transformation Genes (Basel). 2017;8. 37 Tabtabaei S, D'Archivio AA, Maggi MAet al. . Geographical classification of Iranian and Italian saffron sources based on HPLC analysis and UV-Vis spectra of aqueous extracts Eur Food Res Technol. 2019;245:2435-2446.